CLINICAL TRIAL: NCT03766009
Title: Increasing Socioeconomically Disadvantaged Patients' Engagement in Breast Cancer Surgery Decision Making Through a Shared Decision Making Intervention
Brief Title: Increasing Patients' Engagement in Breast Cancer Surgery Decision-Making
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: A231701CD; NCI-2018-00643 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Stage 0; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Institutional cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (surgical consultation) (Active Comparator): Prior to institutional crossover, participants receive care as per usual care.
  Interventions: Other: Usual Care
- Arm II (web-based breast cancer surgery decision aid) (Experimental): Following a 10 week implementation period, at the time of institutional crossover, participants will receive a web-based decision aid prior to the surgical consultation..
  Interventions: Other: Usual Care; Other: Web-based decision aid

INTERVENTIONS:
Other: Usual Care — Usual Care
Other: Web-based decision aid — Web-based decision aid received prior to the surgical consultation
  Arms: Arm II (web-based breast cancer surgery decision aid)

SUMMARY:
This trial studies how well a breast cancer surgery decision aid works in increasing patient engagement in decision making for patients with newly diagnosed stage 0-III breast cancer. The trial also examines barriers to patient engagement even with the use of a decision aid, and if barriers are more likely to be experienced by socioeconomically disadvantaged patients.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. Test the effectiveness of a breast cancer surgery decision aid in increasing patient engagement in decision making (measured by knowledge and power) in clinics serving a high proportion of socioeconomically disadvantaged patients.

II. Test the extent to which the effect of a decision aid on patient engagement is mediated through the mitigation of barriers and determine if persistent barriers are disproportionately experienced by socioeconomically disadvantaged patients.

SECONDARY OBJECTIVES:

I. Characterize how persistent barriers influence patient engagement in decision making in order to identify targets for adjunct interventions that could be implemented in clinics serving a high proportion of socioeconomically disadvantaged patients.

Trial Design:

OUTLINE: This is a multi-site cluster randomized trial using a stepped wedge design. Ten clinics will be recruited for participation. All clinics will begin in the usual care arm. Clinics will be randomized to the timing with which they cross-over to the decision aid intervention, with new clinics crossing over every 10 weeks.

ARM I: usual care

ARM II: decision aid intervention

The only difference between patients enrolled before institutional crossover and patients enrolled after institutional crossover is those who are enrolled after institutional crossover will have been offered the decision aid as accepted practice in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with stage 0-III breast cancer
* Eligible patients must be planning breast surgery as a component of their definitive treatment
* Patients with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss) are not eligible for this study
* Patients with hearing impairment requiring the use of an interpreter are not eligible for this study
* Patients must be able to speak English with the fluency required to have a direct discussion around treatment decision-making (i.e. without interpreter)
* CLINIC STAKEHOLDER (SURGEONS AND CLINIC STAFF): Breast surgeon(s) and nursing staff, medical assistant, or mid-level provider at each participating clinic who participates in the care of patients newly diagnosed with breast cancer
* INSTITUTIONAL: 10 clinics that annually provide surgical care for 120-300 patients newly diagnosed with breast cancer will be selected to participate in this study
* INSTITUTIONAL: Surgeons at eligible clinics must consent to the study as a requirement for site participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2026-12-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Heather B. Neuman,, MD, MS, Study Chair — University of Wisconsin, Madison
Locations (58):
- United States (56):
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam
- Pan American Center for Oncology Trials LLC, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 6 to 12 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
URL: https://www.allianceforclinicaltrialsinoncology.org/main/public/standard.xhtml?path=%2FPublic%2FDatasharing

REFERENCES:
- [Derived] Schumacher JR, Hanlon BM, Zahrieh D, Rathouz PJ, Tucholka JL, McKinney G, Tan AD, Breuer CR, Bailey L, Higham AM, Wecsler JS, Arnold AH, Froix AJ, Dull S, Abbott AM, Fine SG, McGuire KP, Seydel AS, McNamara P, Chow S, Neuman HB. Impact of a Web-Based Decision Aid on Socioeconomically Disadvantaged Patients' Engagement in Breast Surgery Decision-Making: Stepped-Wedge Clinical Trial (Alliance-A231701CD). Ann Surg Oncol. 2025 Aug;32(8):5540-5550. doi: 10.1245/s10434-025-17452-0. Epub 2025 May 17. PMID 40382452
- [Derived] Saucke MC, Jacobson N, McKinney G, Neuman HB. Role of the Surgeon in De-Escalating Emotion During a Breast Cancer Surgery Consultation: A Qualitative Study of Patients' Experiences in Alliance A231701CD. Ann Surg Oncol. 2024 Dec;31(13):8873-8881. doi: 10.1245/s10434-024-16156-1. Epub 2024 Sep 25. PMID 39320397
- [Derived] Zahrieh D, Croghan IT, Inselman JW, Mandrekar SJ. Guidelines for Data and Safety Monitoring in Pragmatic Randomized Clinical Trials Using Case Studies. Mayo Clin Proc. 2023 Nov;98(11):1712-1726. doi: 10.1016/j.mayocp.2023.02.019. PMID 37923529
- [Derived] Schumacher JR, Zahrieh D, Chow S, Taylor J, Wills R, Hanlon BM, Rathouz PJ, Tucholka JL, Neuman HB. Increasing socioeconomically disadvantaged patients' engagement in breast cancer surgery decision-making through a shared decision-making intervention (A231701CD): protocol for a cluster randomised clinical trial. BMJ Open. 2022 Nov 17;12(11):e063895. doi: 10.1136/bmjopen-2022-063895. PMID 36396308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 627 participants were enrolled. Five-hundred and ninety-eight patients (265 UC, 333 DA) were enrolled between June 2019 to December 2021 with 576 (265 UC, 311 DA) during stepped wedge design and 22 extended enrollment beyond Wave 7 (all DA). Twenty-nine surgeons were enrolled between April 2019 to October 2021 with the majority enrolled at the start of the study, while a few additional surgeons were enrolled as they joined the clinic.
Pre-assignment Details: This stepped wedge cluster randomized trial across 10 sites transitioned sites from UC to DA at pre-determined and randomly assigned timepoints, with waves spanning 10-13 weeks each. Sites started in UC and ended with DA. One wave is used for implementation of the DA at the time of crossover, yielding 6 waves for enrollment/data collection.
  The extended enrollment was to enrich the sample for the mixed methods components of the analysis. Surgeon enrollment was not linked to specific wave.
Units Other Than Participants: Sites
Groups:
- Site 1 and 2: 10-13 weeks Usual Care (Participants receive care as per usual care), 10 weeks Implementation (Decision aid implemented at the corresponding clinic) and 65-82 weeks Intervention (Participants receive a web-based decision aid intervention prior to the surgical consultation)
- Sites 3 and 4: 20-26 weeks Usual Care (Participants receive care as per usual care), 10 weeks Implementation (Decision aid implemented at the corresponding clinic), 46-70 weeks Intervention (Participants receive a web-based decision aid intervention prior to the surgical consultation) and 14 Weeks Extended Enrollment Beyond Wave 7 (Participants receive a web-based decision aid intervention prior to the surgical consultation. The extended enrollment was to enrich the sample for the mixed methods components of the analysis.)
- Sites 5 and 6: 56-68 weeks Usual Care (Participants receive care as per usual care), 10 weeks Implementation (Decision aid implemented at the corresponding clinic), 36-39 weeks Intervention (Participants receive a web-based decision aid intervention prior to the surgical consultation) and 1-10 Weeks Extended Enrollment Beyond Wave 7 (Participants receive a web-based decision aid intervention prior to the surgical consultation. The extended enrollment was to enrich the sample for the mixed methods components of the analysis.)
- Sites 7 and 8: 70-71 weeks Usual Care (Participants receive care as per usual care), 10 weeks Implementation (Decision aid implemented at the corresponding clinic), 23-26 weeks Intervention (Participants receive a web-based decision aid intervention prior to the surgical consultation) and 12-15 Weeks Extended Enrollment Beyond Wave 7 (Participants receive a web-based decision aid intervention prior to the surgical consultation. The extended enrollment was to enrich the sample for the mixed methods components of the analysis.)
- Sites 9 and 10: 75-80 weeks Usual Care (Participants receive care as per usual care), 10 weeks Implementation (Decision aid implemented at the corresponding clinic), 10-13 weeks Intervention (Participants receive a web-based decision aid intervention prior to the surgical consultation) and 18 Weeks Extended Enrollment Beyond Wave 7 (Participants receive a web-based decision aid intervention prior to the surgical consultation. The extended enrollment was to enrich the sample for the mixed methods components of the analysis.)
- Surgeons: Surgeons accrual across sites
Period: Usual Care
Arm/Group | Site 1 and 2 | Sites 3 and 4 | Sites 5 and 6 | Sites 7 and 8 | Sites 9 and 10 | Surgeons
Started | 26; 2 Sites | 54; 2 Sites | 34; 2 Sites | 74; 2 Sites | 77; 2 Sites | 28; 10 Sites
Completed | 26; 2 Sites | 51; 2 Sites | 32; 2 Sites | 68; 2 Sites | 76; 2 Sites | 26; 10 Sites
Not Completed | 0; 0 Sites | 3; 0 Sites | 2; 0 Sites | 6; 0 Sites | 1; 0 Sites | 2; 0 Sites
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Treatment goals changed due to metastatic disease | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Transferred care/moved out of state, limited information on chart review | 0 | 1 | 0 | 1 | 0 | 0
Not completed — No treatment or declined surgery | 0 | 0 | 0 | 2 | 0 | 0
Not completed — No surgery but had lymph node dissection instead | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No surgery since patient had a good response to endocrine therapy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other: Staff turnover | 0 | 0 | 0 | 0 | 0 | 2
Period: Implementation
Arm/Group | Site 1 and 2 | Sites 3 and 4 | Sites 5 and 6 | Sites 7 and 8 | Sites 9 and 10 | Surgeons
Started | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 26; 10 Sites
Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 26; 10 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Intervention
Arm/Group | Site 1 and 2 | Sites 3 and 4 | Sites 5 and 6 | Sites 7 and 8 | Sites 9 and 10 | Surgeons
Started | 124; 2 Sites | 109; 2 Sites | 32; 2 Sites | 32; 2 Sites | 14; 2 Sites | 27; 10 Sites
Completed | 118; 2 Sites | 101; 2 Sites | 31; 2 Sites | 25; 2 Sites | 14; 2 Sites | 27; 10 Sites
Not Completed | 6; 0 Sites | 8; 0 Sites | 1; 0 Sites | 7; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Extended Enrollment Beyond Wave 7
Arm/Group | Site 1 and 2 | Sites 3 and 4 | Sites 5 and 6 | Sites 7 and 8 | Sites 9 and 10 | Surgeons
Started | 0; 0 Sites | 16; 2 Sites | 0; 0 Sites | 0; 0 Sites | 6; 2 Sites | 18; 10 Sites
Completed | 0; 0 Sites | 12; 2 Sites | 0; 0 Sites | 0; 0 Sites | 6; 2 Sites | 18; 10 Sites
Not Completed | 0; 0 Sites | 4; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites

BASELINE CHARACTERISTICS:
Population: All stepped-wedge design participants excluding 1 ineligible in UC and 2 refused follow-up at baseline in DA; all extended enrollment beyond wave 7-DA and all surgeons.
Groups:
- UC (Usual Care): Participants receive care as per usual care. Participant assignment to usual care or decision aid intervention was determined by the phase the site was in at time of participant enrollment.
- DA (Decision Aid Intervention): Participants receive a web-based decision aid intervention prior to the surgical consultation. Participant assignment to usual care or decision aid intervention was determined by the phase the site was in at time of participant enrollment.
- Extended Enrollment Beyond Wave 7-DA (Decision Aid Intervention): Participants receive a web-based decision aid intervention prior to the surgical consultation. The extended enrollment was to enrich the sample for the mixed methods components of the analysis.
- Surgeons: Participants consent for participation in site implementation activities, allowing their patients to receive the decision aid, a baseline survey, and audio-recording of their patient consultations.
- Total: Total of all reporting groups
Arm/Group | UC (Usual Care) | DA (Decision Aid Intervention) | Extended Enrollment Beyond Wave 7-DA (Decision Aid Intervention) | Surgeons | Total
Number analyzed (Participants) | 264 | 309 | 22 | 29 | 624
Age, Continuous [Median (Full Range); unit: years] — Population: Age not collected on surgeons
  years
    number analyzed (Participants) | 264 | 309 | 22 | 0 | 595
    (all) | 59 [30 to 87] | 61 [27 to 90] | 63.5 [32 to 84] |  | 61 [27 to 90]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex not collected on surgeons
  Participants
    number analyzed (Participants) | 264 | 309 | 22 | 0 | 595
    Female | 264 | 309 | 22 |  | 595
    Male | 0 | 0 | 0 |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Other includes American Indian or Alaskan Native, Asian, Native Hawaiian or Pacific Islander, Unknown/Not reported for UC, DA, and Extended Enrollment groups; Other includes Asian, Black, and Unknown/Not reported for Surgeons in order to avoid identifying participating surgeons.
  Participants
    Race: White | 169 | 207 | 16 | 18 | 410
    Race: Black | 60 | 62 | 6 | 0 | 128
    Race: Other | 35 | 40 | 0 | 11 | 86
Socioeconomic Disadvantage [Count of Participants; unit: Participants] — Socioeconomic disadvantage was assessed with the Area Deprivation Index measured at the zip+4 level and dichotomized Population: Socioeconomic disadvantage was not collected on surgeons
  Participants
    number analyzed (Participants) | 264 | 309 | 22 | 0 | 595
    Yes | 73 | 59 | 6 |  | 138
    No | 191 | 250 | 16 |  | 457

OUTCOME MEASURES:

1. Primary Outcome: Patient Power: Self-efficacy in Patient Physician Interactions
Description: Power is defined as patients' self-perceived capacity to influence the decision-making encounter. This construct is measured using the Patient's Self-Efficacy in Patient-Physician Interactions (PEPPI)-5 point scale; the primary outcome measure is a total score ranging from 5-25, where higher scores indicate increased self-efficacy. The patient completes the PEPPI-5 questionnaire within 3 weeks post-surgical consultation.
Time Frame: 3 weeks
Population: All stepped wedge design participants who had PEPPI-5 data available excluding 5 UC (1 ineligible, 4 enrolled off-schedule) and 3 DA (2 refused follow-up at baseline, 1 enrolled off-schedule).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | UC (Usual Care) | DA (Decision Aid Intervention)
Number analyzed (Participants) | 238 | 268
score on a scale | 22 [7 to 25] | 22 [5 to 25]

2. Primary Outcome: Patient Power: Active Patient Participation
Description: Power is also separately measured by the validated Active Patient Participation Behaviors System to assess active patient participation during the surgeon consultation and is measured off the audio-recording of the consultation; a summary measure of patient's active involvement in the interaction is coded by the study team and represents a total count of patients' communicative behaviors (i.e., count of patient asking questions, count of patient assertive responses and count of patient expressions of concern) ranging from 0-114, where higher scores indicate increased active patient participation. The consultation for a patient will typically be study day 1 (day of registration).
Time Frame: 1 day
Population: All stepped wedge design participants who had active patient participation behaviors data available excluding 5 UC (1 ineligible and 4 enrolled off-schedule) and 3 DA (2 refused follow-up at baseline and 1 enrolled off-schedule).
Measure: Median (Full Range); unit: count of patient communicative behaviors
Arm/Group | UC (Usual Care) | DA (Decision Aid Intervention)
Number analyzed (Participants) | 258 | 301
count of patient communicative behaviors | 17.5 [0 to 114] | 19 [0 to 112]

3. Secondary Outcome: Patient Knowledge
Description: Patient knowledge is measured from 5 knowledge questions in the Decision Quality Instrument-Breast Surgery survey, with a percent correct recorded as the secondary outcome measure, ranging from 0-100%. The patient completes the Decision Quality Instrument-Breast Surgery survey within 3 weeks post-surgical consultation.
Time Frame: Up to 3 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Concordance Between Personal Values and Surgery Received
Description: This is a binary outcome reflecting whether surgery received (mastectomy; lumpectomy) was concordant or not with the patient's personal values. The patient's personal values are measured from 3 questions on the Decision Quality Instrument (DQI)-Breast Surgery survey; each question ranges from 0 (not at all important) to 10 (extremely important). . The patient completes the DQI within 3 weeks post-consultation. The method by Sepucha et al (2012) will be applied to determine concordance between personal values and surgery received.
Time Frame: Up to 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 827 days
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study for all participants. All-cause mortality was reported for patients through post-operative chart review. All-cause mortality was not reported for surgeons.
Arm/Group | UC (Usual Care) | DA (Decision Aid Intervention)
All-Cause Mortality (participants affected / at risk) | 1/264 | 1/309
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03766009/Prot_SAP_ICF_000.pdf